CLINICAL TRIAL: NCT05754853
Title: An Open-label, Randomized, Multi-center, Phase III Clinical Study of MRG002 Versus Investigator's Choice of Chemotherapy in the Treatment of Patients With HER2-positive Unresectable Locally Advanced or Metastatic Urothelial Cancer Previously Treated With Platinum-based Chemotherapy and PD-1/PD-L1 Inhibitors
Brief Title: A Study of MRG002 Versus Investigator's Choice of Chemotherapy in the Treatment of Patients With HER2-positive Unresectable Advanced or Metastatic Urothelial Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Miracogen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRG002-010
Record Dates: First submitted 2023-02-22; First posted 2023-03-06 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Advanced or Metastatic Urothelium Cancer
Keywords: MRG002; Antibody Drug Conjugate (ADC); HER2; Urothelium Cancer
MeSH Terms: interventions — Docetaxel; Paclitaxel; Gemcitabine; Injections; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MRG002 (Experimental): MRG002 will be administrated by an IV infusion of 2.2 mg/kg on Day 1 of every 3 weeks (21-day cycle).
  Interventions: Drug: Docetaxel Injection; Drug: Paclitaxel Injection; Drug: Gemcitabine Hydrochloride for Injection; Drug: Pemetrexed Disodium Injection
- Docetaxel /Paclitaxel /Gemcitabine Hydrochloride /Pemetrexed Disodium Injection (Active Comparator): Docetaxel injection will be administered by an IV infusion of 75 mg/m2 on Day 1 of every 3 weeks (21-day cycle); Paclitaxel will be administrated by an IV infusion of 175 mg/m2 on Day 1 of every 3 weeks (21-day cycle).
  Gemcitabine Hydrochloride will be administrated by an IV infusion of 1000 mg/m2 on Day 1 and Day 8 of every 3 weeks (21-day cycle).
  Pemetrexed Disodium will be administrated by an IV infusion of 500 mg/m2 on Day 1 of every 3 weeks (21-day cycle).
  Interventions: Drug: MRG002

INTERVENTIONS:
Drug: MRG002 — Administrated intravenously
  Arms: Docetaxel /Paclitaxel /Gemcitabine Hydrochloride /Pemetrexed Disodium Injection
Drug: Docetaxel Injection — Administrated intravenously
  Arms: MRG002
Drug: Paclitaxel Injection — Administrated intravenously
  Arms: MRG002
Drug: Gemcitabine Hydrochloride for Injection — Administrated intravenously
  Arms: MRG002
Drug: Pemetrexed Disodium Injection — Administrated intravenously
  Arms: MRG002

SUMMARY:
The primary objective of this study is to compare the overall survival (OS) and progression-free survival (PFS) between MRG002 and investigator selected chemotherapy in patients with HER2-positive unresectable locally advanced or metastatic urothelial cancer previously treated with platinum-based chemotherapy and PD-1/PD-L1 inhibitors.

DETAILED DESCRIPTION:
This study aims to enroll 290 patients. Participants will be randomly assigned to receive treatment of MRG002 or investigator selected chemotherapy in a 1:1 ratio. The efficacy of MRG002 will be assessed by patient's OS, PFS and other indicators as compared to investigator selected chemotherapy. Additionally, this study will assess the pharmacokinetic profile, immunogenicity, safety, tolerability, and treatment compliance of MRG002.

ELIGIBILITY:
Inclusion Criteria:

* 1. Willing to sign the ICF and follow the requirements specified in the protocol.

  2. Aged 18 to 75 (including 18 and 75), both genders. 3. Expected survival time ≥ 12 weeks. 4. Patients with unresectable locally advanced or metastatic urothelium cancer confirmed by histopathology.

  5. Patients who have failed prior platinum-based chemotherapy and PD-1/PD-L1 inhibitors and have have progressive disease or recurrence on or after their most recent therapy.

  6. Archival or biopsy tumor specimens should be provided (primary or metastatic).

  7. HER2 positive (IHC 3+ or IHC 2+) in the tumor specimens confirmed by central laboratory test.

  8. Patients must have measurable lesions according to the Response Evaluation Criteria in Solid Tumors (RECIST v1.1).

  9. ECOG performance score 0 or 1. 10. Prior anti-tumor treatment-related AEs (NCI-CTCAE v5.0 Criteria) have recovered to ≤ Grade 1 (except alopecia, Grade 2 hypothyroidism, non-clinically significant or asymptomatic laboratory abnormalities).

  11. Organ function must meet the basic requirements. 12. Patients of childbearing potential must take effective contraceptive measures during the treatment and for 180 days after the last dose of treatment.

Exclusion Criteria:

* 1. History of hypersensitivity to any component of MRG002 or history of hypersensitivity of ≥ Grade 3 to trastuzumab.

  2. Patients who have received ADC drugs, or prior taxane, gemcitabine, and pemetrexed for locally advanced or metastatic urothelial cancer; or have received investigational drugs from other clinical trials, chemotherapy, radiotherapy, targeted therapy, or immunotherapy within 4 weeks prior to the first dose; or have received Chinese medicine (herbal medicine) or Chinese patent medicine with anti-tumor indications within 2 weeks prior to the first dose; or have received strong CYP3A4 inhibitors within 2 weeks prior to the first dose or have current requirement of CYP3A4 inhibitors; or had major surgery within 4 weeks prior to the first dose without full recovery or planned surgery within 12 weeks after study treatment.

  3. Patients with clinical symptoms such as plural, abdominal or pericardial effusion requiring puncture drainage.

  4. Patients with central nervous system (CNS) metastasis and/or neoplastic meningitis.

  5. Any severe or uncontrolled systemic diseases. 6. Patients with poorly controlled heart diseases. 7. Evidence of active infections, including but not limited to Hepatitis B, Hepatitis C, or human immunodeficiency virus (HIV) infection.

  8. History of other primary malignancies. 9. History of interstitial pneumonia, severe chronic obstructive pulmonary disease, severe pulmonary insufficiency, symptomatic bronchospasm, etc.

  10. Peripheral neuropathy greater than Grade 1. 11. History of cirrhosis. 12. Patients with active autoimmune disease or a history of autoimmune disease, who are using immunosuppressive agents, or systemic hormone therapy and still receiving them within 2 weeks prior to enrollment.

  13. Uncontrolled tumor-associated bone pain or urgent spinal cord compression. Patients requiring pain control must have been on a stable treatment regimen for at least 2 weeks at the time of first dose 14. Other conditions inappropriate for participation in this clinical trial, at the discretion of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2023-04-06 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Baseline to study completion (up to 36 months)
  OS is defined as the time from the date of randomization until death of any cause.
Progression-Free Survival (PFS) by Independent Review Committee (IRC) | Baseline to study completion (up to 36 months)
  PFS is defined as the duration from the date of randomization to the onset of tumor progression or death of any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Baseline to study completion (up to 36 months)
  ORR is defined as the percentage of patients with a complete response (CR) or partial response (PR) according to RECIST v1.1.
Duration of Response (DoR) | Baseline to study completion (up to 36 months)
  DoR is defined as the time from first documented objective response (CR/PR) to the first onset of tumor progression or death of any nonsurgical cause.
Disease Control Rate (DCR) | Baseline to study completion (up to 36 months)
  DCR is defined as the percentage of patients who achieve CR, PR, and stable disease (SD).
Clinical Benefit Rate (CBR) | Baseline to study completion (up to 36 months)
  CBR is defined as the percentage of patients who achieve CR, PR, and SD for ≥ 6 months.
Time to Response (TTR) | Baseline to study completion (up to 36 months)
  TTR is defined as the duration from randomization to the first documented objective response (CR/PR).
PFS by investigator | Baseline to study completion (up to 36 months)
  PFS is defined as the duration from the date of randomization to the onset of tumor progression or death of any cause.
Adverse Events (AEs) | Baseline to 30 days after the last dose of study treatment
  Any reaction, side effect, or untoward event that occurs during the course of the clinical trial whether or not the event is considered related to the study drug.
Pharmacokinetics (PK) Parameter of MRG002: concentration-time curve | Baseline to 7 days after discontinuation of treatment
  Plot of drug concentration changing with time after drug administration.
Anti-drug antibody (ADA) | Baseline to 7 days after discontinuation of treatment
  The proportion of patients with positive ADA results and its titer.
Neutralizing antibody (NAb) | Baseline to 7 days after discontinuation of treatment
  The proportion of patients with positive NAb results and its titer.

CONTACTS AND LOCATIONS:
Overall Officials: Aiping Zhou, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Fangjian Zhou, MD, Principal Investigator — Sun Yat-sen University Cancer Prevention Center
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No